CLINICAL TRIAL: NCT05599126
Title: A Multicenter Open Study of the Efficacy of Mianserin in Combination With SSRIs in Patients With Depression With Sleep Problems
Brief Title: A Study of Mianserin in Combination With SSRIs in Depression With Sleep Problems
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhenghui YI (Other)
Collaborators: Renhe Tang Pharmaceutical Co. (Unknown); Nantong Mental Health Centre (Nantong Fourth People's Hospital) (Unknown); Brain Hospital of Guangzhou Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Zhenghui YI, Director of Clinical Section VIII, Shanghai Mental Health Center
Organization: Shanghai Mental Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-TX-002
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mianserin; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mianserin with escitalopram (Experimental)
  Interventions: Drug: Mianserin
- Lorazepam with escitalopram (Active Comparator)
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Mianserin — Subjects were required to take mianserin regularly during the study period, with the effective dose being taken orally once a night before bedtime.
  Arms: Mianserin with escitalopram
Drug: Lorazepam — Subjects were required to take lorazepam regularly during the study period, with the effective dose being taken orally once a night before bedtime.
  Arms: Lorazepam with escitalopram

SUMMARY:
Patients with depression with sleep problems have functional abnormalities of 5-HT and NE neurotransmitters, and the NaSSA class antidepressant mianserin has an ameliorative effect on sleep problems along with antidepressant. However, whether mianserin can improve cognitive function in patients still needs to be explored. The benzodiazepine lorazepam can play a central inhibitory role and has good therapeutic effect on insomnia. The mechanism of action of mianserin and lorazepam is different, and there are few comparative studies related to the combination of the two with SSRI drugs for the treatment of depressed patients with sleep problems, and it is unclear whether there are differences in their efficacy and safety. Therefore, to address the above scientific questions, this study was designed to include 100 patients aged 18-60 years with depression with sleep problems, randomly divided into two groups and treated with mianserin + escitalopram or lorazepam + escitalopram, respectively, and followed up for 8 weeks to assess depression and anxiety symptoms, sleep, cognitive function and drug safety. To compare the efficacy and safety of the two regimens in depressed patients with sleep problems and to provide a scientific basis for clinical intervention in depressed patients with sleep problems.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for major depressive disorder (DSM-5) with a HAMD-17 score ≥ 17 and a HAMA score ≥ 14.
* Having complaints of sleep problems or PSQI scores >7.
* Han Chinese, age 18-60 years old, junior high school education or above.
* No previous manic episodes or manifestations of mild manic episodes.
* Not taking antidepressants and sedative-hypnotic drugs in the last 2 weeks, or a 7-day cleansing period for those taking drugs.
* No use of convulsion-free electroconvulsive therapy (MECT) within 8 weeks
* Those who voluntarily participated in the study with the patient's informed consent.

Exclusion Criteria:

* DSM-5 organic mood disorders; psychiatric disorders associated with somatic diseases; psychiatric disorders due to psychoactive substances.
* Those with contraindications to escitalopram, mianserin, lorazepam medications.
* family history of psychiatric or other somatic disorders.
* Those with excessive psychiatric symptoms unable to complete the interview or unable to understand the content of the scale
* Pregnant and lactating females.
* Those who cannot cooperate with the experimental procedure and cannot cooperate effectively.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index,PSQI | 8 weeks
  30% reduction in the PSQI scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided